CLINICAL TRIAL: NCT04121169
Title: Clinical Effectiveness of Egg-derived Polyclonal Antibodies (IM-01) for the Treatment of Mild-moderate Clostridium Difficile Infection (CDI)
Brief Title: Treatment of Mild-moderate Clostridium Difficile Infection (CDI)
Acronym: IM-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmuniMed Inc. (Industry)
Collaborators: University of Calgary (Other); University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-IM-01-2017A; HC6-024-C218566 (Other: Health Canada- Biological and Genetic Therapies Directorate)
Record Dates: First submitted 2019-06-26; First posted 2019-10-09 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-10

CONDITIONS: Clostridium Difficile Infection (CDI)
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Intervention Model Description: Twenty four patients in each group will receive IM-01 treatment at 20g or 10g twice daily:for 10-14 days.
Masking Description: Patients will be randomized 1:1 to receive IM-01 treatment dosage at 20g or 10g twice a day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults subjects with CDI receiving 20g a day (Other): 10 g twice a day for 10 - 14 days
  Interventions: Drug: IM-01
- Adults subjects with CDI receiving 40 g a day (Other): 20 g twice a day for 10 - 14 days
  Interventions: Drug: IM-01

INTERVENTIONS:
Drug: IM-01 — Antibodies react with C. difficile toxin, C. difficile bacteria and spores; neutralizes the toxin and inhibit the growth of spores and vegetative forms of C. difficile
  Other Names: Chicken egg-derived anti-C.difficile polyclonal antibodies

SUMMARY:
Patients diagnosed to have mild-moderate CDI will be randomized to receive IM-01 egg-derived anti-C. difficile polyclonal antibodies in increasing dosages, twice daily, for a total of 10 - 14 days. Resolution of diarrhea and other symptoms and fecal test parameters will be used to assess clinical effectiveness of Immunotherapy with IM-01 antibodies. Patients will be followed for recurrence of CDI. Subjects who are assessed as non-respondents to IM-01 will be reassessed and treated with standard of care CDI antibiotics for 10 -14 days.

DETAILED DESCRIPTION:
INTRODUCTION: BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE The increased incidence of antibiotic resistant 'superbugs' has amplified the use of broad spectrum antibiotics worldwide. An unintended consequence of antimicrobial treatment is disruption of gastrointestinal microbiota, resulting in susceptibility to opportunistic pathogens, such as Clostridium difficile (C. difficile).

C. difficile is a gram-positive, spore-forming, anaerobic bacterium that causes hospital and community-acquired enteric infections resulting in C. difficile-associated diarrhea, pseudo membranous colitis, colitis and death.

Clostridium difficile infection (CDI) remains the predominant cause of health care -associated infectious diarrhea, centered mainly in hospitals but also in the community at a rate of ~100/100,000 population and affecting the elderly disproportionately. Antimicrobial damage to the intestinal microbiome combined with the acquisition of spores of C. difficile is the main cause of pathogenesis. CDI is endemic in hospitals, and although infection control measures have reduced nosocomial rates of CDI in Canada over the past 5 years, community cases now appear to be more apparent .Treatment of CDI utilizes alternate antimicrobials directed at the pathogen, mainly metronidazole, vancomycin, or fidaxomicin given for a recommended 10-14 days. While the majority respond to antibiotic treatment, subsequent recurrences of CDI are observed in 25-40% of patients. Recurrences of CDI are retreated with the same antibiotics and due to the non-selective spectrum of activity of metronidazole and vancomycin, recurrences are increasing in probabilities for subsequent recurrences. Fidaxomicin is relatively more selective and its use is associated with reduced recurrences, but the high cost of fidaxomicin has restricted the usage.

C. difficile infection is a serious diarrheal illness associated with substantial morbidity and mortality and is responsible for hospital and community-acquired diarrhea, pseudo membranous colitis colitis and death..

ImmuniMed Inc. has developed an oral Immunotherapy using egg-derived anti- C. difficile polyclonal antibodies (IM-01), that directly targets the virulence factors of C. difficile. IM-01 is produced from chicken eggs following the immunization of laying hens with C. difficile virulent antigens, C. difficile toxin A, toxin B, C. difficile whole cells and C. difficile spores. IM-01 is in the form of spray-dried whole egg powder (yolk plus egg white containing ovalbumin) and is very stable for functional activity. Upon reconstitution, IM-01 is administered orally, which allows it to reach to the intestinal lumen, where C. difficile toxins exert their toxic effects. In addition, IM-01 antibodies bind to C. difficile toxins and spores and neutralize their biological activities in vitro.

The use of polyclonal antibodies derived from chicken eggs (IgY) to confer passive immunity has gained attention as a novel strategy for oral immunotherapy as an alternative to antibiotics for treatment of intestinal pathogens which cause diarrhea in animals and humans including, enterotoxigenic E. coli, Salmonella spp, and both bovine and human rotaviruses. Compared with mammalian antibodies (IgG), chicken egg-derived antibodies (IgY) have high antigen-specificity and avidity, react more rapidly to the same antigens and differ from mammalian antibodies (IgG) in both structural and immunological properties.. Compared to IgG, IgY is more stable in gut at pH 3.5 -11 and better tolerates enzymatic degradation by trypsin and chymotrypsin; the stability of IgY against pepsin is pH-dependent.

Immunimed has determined that IgY polyclonal antibodies-specific to E. coli in egg powder containing albumin, are functionally stable when stored at 2-8°C for over 10 years.

This makes IM-01 antibodies attractive for oral immunotherapy since eggs are normal dietary components, with no known toxic side effects. The IM-01 antibodies are shown to bind with C. difficile toxins and spores as well as to neutralize their biological activities in vitro.

Compared with active vaccination, passive immunotherapy using IM-01 egg-derived polyclonal anti-C. difficile antibodies has advantages including: (i) rapid and local onset of action, (ii) highly specific activity, (iii) applicability to a broader range of patients from children to adults including immunocompromised patients, (iv) strategically can be applied for a specific event when it occurs, in contrast to a vaccination model where large populations need to be treated in advance and sustain active antibodies for long-durations, and (v) is a normal part of human diet.

In a published literature, hamsters treated orally with C. difficile anti-toxin A and anti-toxin B neutralizing egg-derived polyclonal antibodies were protected following C. difficile challenge. Also, hamsters treated with egg-derived antibodies did not develop relapsing disease months after the treatment with antibodies. .

Furthermore, egg-derived polyclonal antibodies have several advantages over the monoclonal antibodies (MAbs), since MAbs are generally specific for single epitope, when polyclonal antibodies - a new class of biopharmaceuticals, that have higher affinities for multiple target antigens and can recognize multiple epitopes resulting in superior potency; since they can recognize multiple toxin epitopes as it is relevant to polymorphism of the toxin A and toxin B genes in C. difficile.

A piglet study was performed to demonstrate the safety and therapeutic effect of egg-derived polyclonal antibodies -specific to E. coli K-88, in farm animals. It has been established that E. coli K88 that cause diarrhea in piglets by colonizing in the lower GI tract of piglets improve their growth performance following treatment with E. coli K-88-specific antibodies orally.Furthermore, the highest body weight gain was achieved in pigs which were fed with the highest dosage of E. coli K-88 antibodies (4kg/1000 kg of nursery diet) compared to the lowest antibody dosage (1kg /1000 kg of nursery diet).

It was concluded that feeding of piglets with egg-derived polyclonal antibodies-specific to E. coli K-88 results in significantly improved growth performance in an antibody dose-dependent manner. The manufacturing process for egg-derived polyclonal antibodies targeted to enterotoxigenic E. coli has been approved and validated by the Canadian Center for Veterinary Biologics.

In conclusion oral Immunotherapy using polyclonal antibodies is considered to have a high safety profile with a low likelihood of adverse effects. If proven to be effective as an anti-infective approach, antibiotic selection pressure could be reduced, a key strategy to limit antibiotic resistance in C. difficile infections.

IM-01 is spray-dried egg powder product containing polyclonal antibodies -specific to C. difficile toxins A and toxin B, plus antibodies to C, difficile spores. A 20g/day dosage of IM-01 was selected based on a pre-clinical animal study data, using piglets to treat with C. difficile enteritis.disease with 0.6g of IM-01 orally daily for 4 days.

Under compassionate grounds, patients with confirmed CDI clinical diagnosis with unformed diarrheal stools, abdominal cramps and a positive stool test for the presence of toxins and/or C. difficile in culture, 106 patients (ages: 11-93 years) were enrolled for the clinical study. All patients signed informed consent forms to participate in the study. The amount of IM-01 antibody powder product (10g or 20g) orally administered daily by each patient with 150 mL of milk and followed for up to 6-week period following IM-01 immunotherapy. Seventy six patients received an oral dose of 20 g of IM-01 and 30 patients received 10 g of IM-01 powder daily for 10 consecutive days, as drinkable therapy with milk or chocolate milk. The primary endpoint of the study was to eradicate C. difficile in stool samples.

Of the 106 patients treated with IM-01 therapy,101 patients showed significant improvement of clinical symptoms with negative stool test results for CDI.Five patients showed reduced clinical symptoms during IM-01 treatment period. No recurrence was observed with IM-01 therapy during the follow up period. No safety concerns were reported.

Standard of care (SOC) antibiotics for the treatment of CDI have observed responses to treatment i.e. resolution of diarrhea and ancillary symptoms/signs in 72-88% of subjects, and for those subjects who do achieve resolution of CDI, ~16-24% experience a recurrence of CDI within an 8 week follow up. Non-responders are treated with higher dosages of vancomycin. day interval. A post-treatment minimal follow up period of 30 days has been used in recent RCTs of antimicrobials. Other trials have used several time points i.e 8 weeks or 12 weeks post -treatment. Therefore, in absence of a standard of care control arm, the foregoing response rates for resolution of CDI symptoms (~80%), and a recurrence rate of 20% will be used for as a response template for this study. In the absence of randomization of subjects to an antibiotic treatment control group,

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged 18 to 89
* In good general health as evidenced by medical history or Diagnosed with specific condition/disease or Exhibits specific clinical signs or symptoms or physical/oral examination findings
* Participant has a diagnosis of CDI defined as (i) presence of diarrhea with 4 or more unformed stools within 24 hours and (ii) positive test for toxigenic C. difficile from stools collected within 7 days.
* Participants received < 24 h of SOC therapy for CDI.
* Participants presented with primary CDI episode or any number of CDI relapse recurrence of CDI
* Participants comply with the eligibility criteria and willing to participate in the study including the 8 week post treatment follow up period.
* White Blood Cell absolute neutrophil count <15 x 109/L,
* Women of reproductive potential must use highly effective contraception. For those with child bearing potential, the following methods of birth control are required from Visit 1 up to at least 30 days after study treatment discontinuation: 1). Diaphragm, female condom or cervical cap, partner's use of a condom, any of which must be used in combination with a spermicide; 2). Intra-uterine device; 3). Oral or injectable contraceptive agent, implant, or transdermal contraceptive hormone patches. If a hormonal contraceptive is used, it must have been taken for at least one month prior to enrolment/randomization; 4). Sterilization method (tubal ligation/occlusion, or partner's vasectomy); 5). True abstinence from intercourse with a male partner only when this is in line with the preferred lifestyle of the subject.
* Men of reproductive potential must use condoms-

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* known allergic reactions to chicken egg components.
* Female of child bearing potential and not receiving contraception; pregnant or lactating persons.
* severe CDI defined as >10 unformed bowel movements (UBMs)/24 h period, fever >38.5 o C, White Blood Cell count > 15 x 109/L, abdominal pain and tenderness on physical examination, toxic megacolon, ileus, nausea, vomiting.
* receipt of > 24 h of SOC treatment of CDI, or fecal microbial transplant (FMT) prior to enrollment.
* treatment with another investigational drug or other intervention within 30 days prior to enrollment including intravenous immunoglobulin (IVIG) or monoclonal intravenous (IV) antibody.
* received vaccine for C. difficile.
* concurrent use of probiotics of any type during treatment and follow up.
* unable to discontinue use of opiates for diarrhea control.
* co-infection with another gastrointestinal (GI) pathogen.
* presence of Inflammatory Bowel Disease (IBS), IBS with diarrhea (IBS-D), chronic diarrhea of unknown cause.
* any condition that hinders oral consumption. Exception: nasogastric tubes can be used to administer the product.
* death likely within study interval.
* any circumstance or medical condition under the Investigator's opinion that precludes participation.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or Female
Enrollment: 60 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Determine Clinical Response to IM-01 Treatment for CDI for 14 days | 10-14 days of IM-01 post-treatment
  Decrease the frequency of unformed bowel motions to less than 3 per day and sustain for the duration of treatment to 10-14 days.
Reduce C. difficile pathogen count, spore count, and C. difficile Toxin Titers in stool samples following IM-01 treatment, | day 56 IM-01 post-treatment
  To enumerate numbers of C.difficile present per g of stool by dilution at plate counts on CCFA or Biomerieux C. difficile Chrom Agar , Total counts on three plates express as log 10 count /g versus spore counts after alcohol shock. Toxin titers: expressed as 1/dilution of the fecale filtrate neutralized by specific anti-toxin antibodies from Tech Lab using the CCNA test. .

SECONDARY OUTCOMES:
Rate of recurrence of CDI in day 44, day 56 and day 70 IM-01 post-treatment follow up period | day 44, 56 and 70 post- IM-01 treatment
  In those that responded to treatment with resolution of CDI, the rate of recurrence of CDI in a 30, 42 and 56 day follow up period.
  • Exploratory outcome: patterns of C. difficile microbial counts and toxin titres in relationship to clinical outcomes from treatment assignments

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Louie, MD,FRCPC, Principal Investigator — University of Calgary Foothills Medical Center
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] LITERATURE REFERENCES 1. Halsey J. Am. J. Health-Syst Pharm 65: 705-715, 2008. 2. Lessa, F.C et al. N.Eng.J.Med.372: 825-834, 2015. 3. Kee, V. R. Amer. J. Geriatric Pharmacotherapy. 10: 14-24, 2012 4. Centers for Disease Control and Prevention. Vital signs: Making healthcare safer. Stopping C. difficile infections. http:/www.cdc.gov/vitalsigns/Hai/StoppingC.difficile/. March, 2012 5. Comparison of the burdens of hospital-onset, healthcare facility-associated Clostridium difficile Infection and of healthcare-associated infection due to methicillin-resistant Staphylococcus aureus in community hospitals. Miller B.A. et al. Infect Control Hosp Epidemiol. 32:387-390, 2011. 6. (APIC) National Prevalence study for Clostridium difficile in US Healthcare Facilities. November 11, 2008. 7. European Society of Clinical Microbiology and Infectious Diseases (ESCMID): treatment guidance document for Clostridium difficile infection (CDI). Bauer , M.P.; Kuijper, E.J. van Dissel, I.T;. Clin. Microbiol. Infect. 2009, 15: 1067-79. 8. Society for Healthcare Epidemiology of America; Infectious Disease Society of America Clinical Practice guidelines for Clostridium difficile infection in adults: 2010 updates by the Society for Healthcare Epidemiology of America (SHEA) and the Infectious Disease Society of America (IDSA). Cohen S.F.; Gerding, D.N.; Johnson, S; et al. Infect. Control Hosp. Epidemiol. 2010, 31: 431-55. 9. Treatment of First recurrence of Clostridium difficile Infection Fidaxomicin Versus Vancomycin. Cornely, O.A; Miller, M.A; Louie, T.J. et al. Clin. Infect. Dis. 2012, 55 (Suppl 2) S154-61. 10. Fidaxomycin versus Vancomycin for C. difficile infections. Louie, T.J; Miller, M.A.; Mullane. D.O et al. New Eng. J. Med. 2011, 364: 422031. 11. Consequence of Clostridium difficile infection: Understanding of healthcare burden. Bouza E. Clin. Microbiol. Infect. 18 (suppl 6) 5-12, Dec 2012. 12. Emergence and global spread of epidemic healthcare-associated Clostridium difficile. He M, Miyajima F, Roberts P et al. Nat. Genet. 45: 109-113, 2012. 13. PCR ribotyping and antimicrobial susceptibility testing of isolates of Clostridium difficile cultured from toxin-positive diarrheal stools of patients receiving medical care in Canadian hospitals: the Canadian Clostridium difficile Surveillance Study (CAN-DIFF) 2013-2015. Karlowsky J. A et al. Diag. Microbiol and Infect Dis. Vol 91. Pages 105-111, 2018 . 14. Antibodies for Treatment of Clostridium difficile Infections. Humphreys, D.P. and Wilcox, M.H. Clinical and Vaccine Immunology 21: 913-923, 2014. 15. Association between antibody response to toxin A and protection against recurrent C. difficile diarrhea. Kyne l et al. Lancet 357: 189-193, 2001. 16. IgG Antibody Response to Toxin A and Toxin B in patients with Clostridium difficile Infection. Wullt M et al. Clin. Vaccine Immunol. 19; 1552-54, 2012. Protocol CP-IM-01-2017A 10 July 2018 (Version 5) ________________________________________________________________________________________________________